CLINICAL TRIAL: NCT07008703
Title: Phase Ib/IIa Clinical Trial to Evaluate the Safety, Efficacy, and Pharmacokinetic Characteristics of SSS40 in Subjects With Moderate to Severe Bone Metastasis Cancer Pain
Brief Title: Phase I Study of sss40 Injection for Moderate-to-Severe Bone Metastatic Cancer Pain
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSS-SSS40-MBP-I-02
Record Dates: First submitted 2024-01-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain | interventions — Nerve Growth Factor; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SSS40 (Experimental): Drug: Injection of humanized nerve growth factor (NGF) antibody， Dosage Form: Injection， Dosage: 20-60 mg ， Frequency: Single dose， Duration: efficacy assessed over 12 weeks
  Interventions: Drug: Injection of humanized nerve growth factor (NGF) antibody

INTERVENTIONS:
Drug: Injection of humanized nerve growth factor (NGF) antibody — Subcutaneous injection, 20mg
  Other Names: SSS40

SUMMARY:
This is a Phase Ib/IIa, multicenter, sequential clinical trial evaluating the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of SSS40 injection in patients with moderate-to-severe bone metastatic cancer pain. The study includes two stages: a single-arm, open-label, dose-escalation and dose-expansion Phase Ib followed by a randomized, double-blind, placebo-controlled Phase IIa.

DETAILED DESCRIPTION:
The study consists of two sequential phases:

Phase Ib - Dose-Escalation and Dose-Expansion:

This phase is a single-arm, multicenter, open-label clinical trial involving single-dose administration of SSS40 injection. Patients will be enrolled into sequential dose cohorts to evaluate the safety, tolerability, and PK profile of escalating doses of SSS40. Based on observed adverse events, particularly dose-limiting toxicities (DLTs), and PK data, the sponsor and investigators will determine whether adjustments to the dose escalation scheme (e.g., dosing interval, cohort size) are needed or if additional unplanned dose levels should be added. Following initial dose-escalation, a dose-expansion cohort will be conducted at the selected dose level to further characterize safety and gather additional preliminary efficacy data.

Phase IIa - Randomized, Double-Blind, Placebo-Controlled Trial:

After sufficient safety and efficacy data are obtained from Phase Ib, the sponsor and investigators may proceed to Phase IIa. This phase will be a randomized, double-blind, placebo-controlled study designed to further assess the efficacy, safety, tolerability, immunogenicity, and PK of SSS40 injection in patients with moderate-to-severe bone metastatic cancer pain. Patients will be randomly assigned to receive either SSS40 injection or placebo, and outcomes including pain intensity, analgesic use, and quality of life measures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily sign an informed consent form, voluntarily participate in the trial, and are willing and able to receive medication, examination, visits, and other related operations according to the trial protocol;
2. When signing the informed consent form, adult male or female subjects aged ≥ 18 years old；
3. Previous medical records confirm that the subject has cancer and is diagnosed with bone metastasis; During screening or within 120 days prior to screening visits, Confirming bone metastasis through imaging according to local medical standards, such as bone scans, magnetic resonance imaging (MRI), computed tomography (CT) scans, or positron emission computed tomography (PET-CT) Scanning, diagnosed as bone metastasis based on CT/MRI/PET-CT. If the above examination is not performed within 120 days, a bone scan confirmation is required. If imaging only involves bone scanning, additional CT, MRI, or PET is required to confirm bone metastasis；
4. Weight ≥ 40kg during screening；
5. Expected survival time ≥ 3 months；
6. Pain at the site of cancer bone metastasis, with an average pain score of ≥ 4 points at the designated pain point of bone metastasis (screening period and baseline evaluation period of 3 days)；
7. When screening, the Eastern Oncology Collaborative Group (ECOG) physical condition score was ≤ 2 points；
8. The subjects are willing not to use prohibited drugs throughout the entire study period；
9. The subjects are willing to refrain from using chemotherapy drugs with significant bone marrow suppression from 14 days before administration to 28 days after administration. Among them, drugs with significant bone marrow suppression include paclitaxel (PTX), docetaxel (TXT), vinorelbine (NVB), tiniposide (VM-26), vindesin (VDS), etoposide (VP-16), carboplatin (CBP), mitoxantrone (MITX), nitrogen mustard (HN2), daunorubicin (DNR), and doxorubicin (ADM) [THP, MTX, 6-MP, and IFO]；
10. During screening, the bone marrow function of the subjects meets the following requirements (if necessary, can be repeated for confirmation): a. Absolute neutrophil count (ANC) ≥ 1500/mm3 or ≥ 1.5 × 109/L; b. Platelet count ≥ 90000/mm3 or ≥ 90 × 109/L; c. Hemoglobin ≥ 70.0 g/L；
11. When screening, the renal function meets the following requirements (if necessary, repeat the examination to confirm): a Estimated glomerular filtration rate ≥ 30 mL/min, and b. Urinary protein<2+；
12. During screening, liver function meets the following requirements (if necessary, can be repeated for confirmation): a. Total serum bilirubin ≤ 1.5 × ULN; b. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5.0 if the tumor affects the liver) × ULN; c. Alkaline phosphatase ≤ 5 × ULN；
13. If the subject is not currently receiving anticoagulant therapy, the international standardized ratio (INR) or prothrombin time (PT) during screening should be less than 1.5 × ULN (can be double checked to confirm if necessary). Subjects currently receiving anticoagulant therapy must have an INR within the recommended range applicable to their clinical status；
14. Female participants of childbearing age must agree to use reliable contraceptive measures within 6 months after the start of the study medication and have no plans to conceive or donate eggs; Male participants must agree to use reliable contraceptive measures within 6 months of starting the study medication and have no plans for childbirth or sperm donation；
15. The subjects are able to communicate well with the researchers and complete the study in accordance with the research regulations.

Exclusion Criteria:

1. During screening, there was hypercalcemia (blood calcium concentration ≥ 2.75mmol/L or 11.0mg/dL)；
2. The pain of the subjects is caused by reasons unrelated to cancer bone metastasis (such as intestinal obstruction/perforation, spinal cord compression, brain metastasis, pathological fractures or near fractures, etc.)；
3. The pain of the subjects is neuropathic pain, visceral pain, or unknown in nature, caused by previous anti-tumor treatment, infection, or other reasons mainly unrelated to bone metastasis；
4. Subjects with brain or meningeal metastases (patients with stable brain metastases can be included in this study)；
5. Starting systemic treatment for primary malignant tumors or bone metastases within 14 days prior to the first day of the baseline assessment period, including chemotherapy and hormone therapy (excluding those who have received stable treatment for at least 30 days prior to the first day of the baseline assessment period and still meet the inclusion criteria for bone pain severity)；
6. Individuals who have developed peripheral neuropathy and unstable neuropathy after receiving radiation therapy for bone metastases within 30 days prior to the first day of the baseline evaluation period；
7. Individuals who receive unstable radiation therapy within 30 days prior to the first day of the baseline evaluation period or experience a significant decrease in NRS score (by more than 3 points) after radiation therapy；
8. Starting within 30 days prior to the baseline evaluation period, unstable doses of adjuvant analgesic therapy (such as unstable doses combined with single agent acetaminophen (paracetamol), serotonin/norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, antiepileptics, bisphosphonates, desukumab, corticosteroids or muscle relaxants, etc.) should be used；
9. Diagnosed as knee or hip arthritis or Kellgren Lawrence grade ≥ 2 according to the American Rheumatology Association (ACR) and clinical and imaging standards；
10. Screening for major injuries or surgeries in major joints (such as hip, knee, or shoulder) within the previous year; Individuals with a history of osteonecrosis or osteoporotic fractures (i.e., subjects with osteoporosis and mild traumatic or non traumatic fractures) or a history of joint related events, such as meniscus or knee ligament injuries (with or without surgical repair) or joint infections；
11. Imaging atlas, determined by researchers, with imaging evidence indicating any of the following diseases during screening: a) rapidly progressive osteoarthritis, b) atrophic or malnourished osteoarthritis, c) subchondral incomplete fractures, d) spontaneous knee joint osteonecrosis (SPONK), e) osteonecrosis, f) pathological fractures, g) neuroarthritis (Charcot's joint), h) crystalline arthritis, i) rheumatoid arthritis, j) lupus erythematosus, k) Significant knee joint effusion or active infection, l) shoulder osteoarthritis and other diseases. Note: i. Patients with bone necrosis secondary to radiotherapy (i.e. radiation-induced osteonecrosis) and related to bone metastasis (i.e. involving the tumor bone interface) are allowed to participate in this study. Ii. Subjects with pathological vertebral fractures with vertebral body damage less than 50% and no spinal canal damage are allowed to participate in this study. Iii. Subjects with pathological fractures of non weight-bearing bone (such as humerus) that have been treated (such as fixation) and have healed, if the fracture does not involve the large joint, can participate in this study；
12. Individuals with a clinically significant history of heart disease, including those classified by the New York Heart Association as grade III or IV congestive heart failure, left ventricular insufficiency ejection fraction<35%, ischemic heart disease, surgical treatment for coronary artery disease, and significantly abnormal electrocardiograms (resting tachycardia (heart rate ≥ 120 beats/min) or resting bradycardia (heart rate ≤ 45 beats/min) within the first 6 months of screening；
13. Diagnosed as transient ischemic attack or stroke with sequelae (such as aphasia, significant motor or sensory dysfunction) within the first 6 months of screening；
14. A clinically significant history, diagnosis, or symptoms and signs of neurological diseases, including but not limited to: a Alzheimer's disease or other types of dementia; b. Head trauma with clinical significance within the past year; c. Peripheral neuropathy or autonomic neuropathy (including chemotherapy related peripheral neuropathy); d. Epilepsy or epilepsy related diseases, with a history of epileptic seizures within 2 years prior to screening; e. Myopathy；
15. Individuals with an overall impact score greater than 7 on the Autonomous Neurological Symptom Survey (SAS) during screening；
16. Individuals with a history of carpal tunnel syndrome (CTS) and experiencing symptoms or signs of CTS within the year prior to screening；
17. Individuals with a history of allergic reactions or rapid allergic reactions to therapeutic or diagnostic monoclonal antibodies or IgG fusion proteins；
18. Positive cases of active hepatitis, HIV infection, and Treponema pallidum infection were found during screening；
19. Vaccination received one month before screening；
20. Screening for individuals with a significant history of alcohol abuse, abuse of analgesics or anesthetics within the first 6 months (excluding medications currently under treatment)；
21. Previous exposure to exogenous nerve growth factor or anti nerve growth factor antibodies；
22. Participate in other clinical studies within 30 days prior to the baseline evaluation period (90 days for investigational biologics)；
23. The presence of severe acute or chronic diseases, mental disorders, or laboratory test abnormalities may increase the risk of subjects participating in this study or receiving treatment with study drugs, or may affect the interpretation of the research results. According to the judgment of the researchers, these conditions may make the subjects unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) Events (NCI-CTCAE V5.0) | Up to Day 85
  All adverse events occurring during the entire study period will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE Version 5.0)

SECONDARY OUTCOMES:
Pain intensity maximum change from baseline (NRS) | Week 12
  The mean change in Numerical Rating Scale (NRS) pain score from baseline within 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shuxia Luo, Principal Investigator — HenanCancerHospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No